CLINICAL TRIAL: NCT05139875
Title: A Comparative Study of Betamethasone (Diprospan) and Triamcinolone Acetonide as Single Intra-Articular Injection in Knee Osteoarthritis, A Double-Blinded, Randomized Controlled Trial
Brief Title: Comparing Intra-articular Betamethasone (Diprospan) and Triamcinolone Acetonide Injection in Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Kittipong Wattanasirisombat, Principal investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTU-EC-OT-1-266/64
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
Keywords: Intra-articular injections; Corticosteroids; Triamcinolone acetonide; Betamethasone; Nonoperative management
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — betamethasone-17,21-dipropionate; betamethasone sodium phosphate; betamethasone dipropionate, betamethasone sodium phosphate drug combination; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Participants are randomized and assigned to betamethasone (Diprospan) group or Triamcinolone acetonide group in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 1. Participant and Care Provider will not know which drug is injected to the investigated knee because the opaque syringe is used to inject.
  2. Investigator and outcomes assessor will not known the group of participants because randomization, they only know the number of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Betamethasone (Diprospan) (Experimental): Participant received single intra-articular Betamethasone Dipropionate / Betamethasone Sodium Phosphate 1 ml
  Interventions: Drug: Betamethasone Dipropionate / Betamethasone Sodium Phosphate
- Triamcinolone acetonide (Active Comparator): Participant received single intra-articular Triamcinolone acetonide 40 mg
  Interventions: Drug: Triamcinolone Acetonide 40mg/mL

INTERVENTIONS:
Drug: Betamethasone Dipropionate / Betamethasone Sodium Phosphate — Single intra-articular Betamethasone Dipropionate / Betamethasone Sodium Phosphate (Diprospan) injections to affected knee
  Other Names: Diprospan
  Arms: Betamethasone (Diprospan)
Drug: Triamcinolone Acetonide 40mg/mL — Single intra-articular Triamcinolone Acetonide injections to affected knee
  Other Names: Kanolone-F
  Arms: Triamcinolone acetonide

SUMMARY:
The purpose of this study is to compare the efficacy of Intra-articular corticosteroid injection between Betamethasone (Diprospan) and Triamcinolone acetonide for treatment of knee osteoarthritis

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be chosen for eligibility for the study entry. At day 0 (before intra-articular injection), patients who meet the eligibility criteria will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to Betamethasone (Diprospan 1 ml) or Triamcinolone acetonide (40 mg) single intra-articular injection

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic Primary knee osteoarthritis (Kellgren-Lawrence stage 2 or 3)
2. Failed other conservative treatment
3. Comply with protocol

Exclusion Criteria:

1. Allergy to any of the medications in this protocol (Betamethasone, Triamcinolone, Paracetamol, Tramadol)
2. Previous fracture or surgical procedure
3. Previous intra-articular injection in the past 6 months
4. Previous oral Symptomatic slow-acting drugs for osteoarthritis (SYSADOA) (Glucosamine, Diacerein) used in the past 6 months
5. Current infection in the affected limb
6. Uncontrolled Diabetes Mellitus
7. Primary or secondary adrenal insufficiency
8. Coagulopathy or current anticoagulant used
9. Current steroid used
10. Lower extremity weakness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Difference of 100-mm Visual analog scale (VAS) Pain Score between Betamethasone (Diprospan) and Triamcinolone group | Baseline before intra-articular injection, 1 day, 2 days, 3 days, 1 week, 3 weeks, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months after the day of intra-articular injection
  * The 100-mm VAS pain score is a self-reported instrument assessing Pain Score at 1 day, 2 days, 3 days, 1 week, 3 weeks, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months after the day of intra-articular injection
  * Participants will assess the VAS pain score at rest and on-movement
  * VAS Pain at rest is evaluated when the participant's wakeup in the morning
  * VAS Pain on-movement is evaluated when the participant's walking for 10 meters and then resting for 5 minutes
  * Possible scores range from 0 (no pain) to 100 (worst imaginable pain)
  * Higher scores mean a worse pain

SECONDARY OUTCOMES:
Difference of Modified Western Ontario and McMaster Universities Arthritis Index (WOMAC) score between Betamethasone (Diprospan) and Triamcinolone group | Baseline before intra-articular injection,1 month, 3 months, 6 months after intra-articular injection
  * The Modified WOMAC score is a validated, self-reported instrument consisting of 24 items divided into 3 subscales (Pain, Stiffness, Physical function).
  * The test questions are scored on a scale of 0-4, which corresponds to None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  * Possible scores range from 0-20 for pain, 0-8 for Stiffness, 0-68 for Physical function.
  * a sum of the scores for all three subscales gives a total WOMAC score (0-96)
  * Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Difference of University of California and Los Angeles (UCLA) score between Betamethasone (Diprospan) and Triamcinolone group | Baseline before intra-articular injection,1 month, 3 months, 6 months after intra-articular injection
  * The UCLA is a 10-point scale measurement that evaluates patients' daily activity levels.
  * The 10-point scale is leveled from 1 to 10 (1= worst, 10 = best).
  * Level 1 is wholly inactive and dependent on others, while level 6 is unlimited housework and shopping and level 10 is regular participation in impact sports, such as jogging or tennis.
Difference of Range of motion between Betamethasone (Diprospan) and Triamcinolone group | Baseline before intra-articular injection,1 month, 3 months, 6 months after intra-articular injection
  - Flexion and extension angle of the knee is measured by a long-arm goniometer
Difference of Time up-and-go test between Betamethasone (Diprospan) and Triamcinolone group | Baseline before intra-articular injection,1 month, 3 months, 6 months after intra-articular injection
  * The Time up-and-go test (TUGT) measures the time (seconds) that the patient takes to rise from a chair and walk for 3 meters. Then, he or she turns around and comes back to the seat at the initial position.
  * They were permitted to use walking aids if they wished.
  * TUGT was a reliable and valid test for quantifying functional mobility.
Difference of 2-minutes walking test between Betamethasone (Diprospan) and Triamcinolone group | Baseline before intra-articular injection,1 month, 3 months, 6 months after intra-articular injection
  * Participants were instructed to walk for 2 minutes at their normal pace up and down a designated corridor, turning around at each end of the corridor without stopping
  * They were permitted to use walking aids if they wished.
  * The results were recorded as the total distance walked in meters.
Incidence of side effects of intra-articular steroid injection | 1 month, 3 months, 6 months after intra-articular injection
  Injection site reaction, Erythema, Swelling, Injection-site pain, Pruritus, cellulitis were observed after intra-articular injection.
Difference of Total Paracetamol and Tramadol used between Betamethasone (Diprospan) and Triamcinolone group | 6 months after intra-articular injection
  * Post-injection protocol, Participants can use Paracetamol 500 mg 2 tabs every 4 hours for knee pain if it did not relieve the pain they can take Tramadol 50 mg 1 cap every 6 hours.
  * The total use of Paracetamol and Tramadol was recorded. (tablet)

CONTACTS AND LOCATIONS:
Overall Officials: KITTIPONG WATTANASIRISOMBAT, MD, Study Director — Thammasat University
Locations (1):
- Thammasat University Hospital, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Background] Uson J, Rodriguez-Garcia SC, Castellanos-Moreira R, O'Neill TW, Doherty M, Boesen M, Pandit H, Moller Parera I, Vardanyan V, Terslev L, Kampen WU, D'Agostino MA, Berenbaum F, Nikiphorou E, Pitsillidou IA, de la Torre-Aboki J, Carmona L, Naredo E. EULAR recommendations for intra-articular therapies. Ann Rheum Dis. 2021 Oct;80(10):1299-1305. doi: 10.1136/annrheumdis-2021-220266. Epub 2021 May 25. PMID 34035002
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Rheumatol. 2020 Feb;72(2):220-233. doi: 10.1002/art.41142. Epub 2020 Jan 6. PMID 31908163
- [Background] Jevsevar DS, Brown GA, Jones DL, Matzkin EG, Manner PA, Mooar P, Schousboe JT, Stovitz S, Sanders JO, Bozic KJ, Goldberg MJ, Martin WR 3rd, Cummins DS, Donnelly P, Woznica A, Gross L; American Academy of Orthopaedic Surgeons. The American Academy of Orthopaedic Surgeons evidence-based guideline on: treatment of osteoarthritis of the knee, 2nd edition. J Bone Joint Surg Am. 2013 Oct 16;95(20):1885-6. doi: 10.2106/00004623-201310160-00010. No abstract available. PMID 24288804
- [Background] Oo WM, Liu X, Hunter DJ. Pharmacodynamics, efficacy, safety and administration of intra-articular therapies for knee osteoarthritis. Expert Opin Drug Metab Toxicol. 2019 Dec;15(12):1021-1032. doi: 10.1080/17425255.2019.1691997. Epub 2019 Nov 13. PMID 31709838
- [Background] Garg N, Perry L, Deodhar A. Intra-articular and soft tissue injections, a systematic review of relative efficacy of various corticosteroids. Clin Rheumatol. 2014 Dec;33(12):1695-706. doi: 10.1007/s10067-014-2572-8. Epub 2014 Mar 21. PMID 24651914
- [Result] Douglas RJ. Corticosteroid injection into the osteoarthritic knee: drug selection, dose, and injection frequency. Int J Clin Pract. 2012 Jul;66(7):699-704. doi: 10.1111/j.1742-1241.2012.02963.x. PMID 22698422
- [Result] Cole BJ, Schumacher HR Jr. Injectable corticosteroids in modern practice. J Am Acad Orthop Surg. 2005 Jan-Feb;13(1):37-46. doi: 10.5435/00124635-200501000-00006. PMID 15712981
- [Result] Schumacher HR, Chen LX. Injectable corticosteroids in treatment of arthritis of the knee. Am J Med. 2005 Nov;118(11):1208-14. doi: 10.1016/j.amjmed.2005.05.003. PMID 16271901
- [Result] Husby G, Kass E, Spongsveen KL. Comparative double-blind trial of intra-articular injections of two long-acting forms of betamethasone. Scand J Rheumatol. 1975;4(3):118-20. doi: 10.3109/03009747509165439. PMID 1101375
- [Result] Liu D, Ahmet A, Ward L, Krishnamoorthy P, Mandelcorn ED, Leigh R, Brown JP, Cohen A, Kim H. A practical guide to the monitoring and management of the complications of systemic corticosteroid therapy. Allergy Asthma Clin Immunol. 2013 Aug 15;9(1):30. doi: 10.1186/1710-1492-9-30. PMID 23947590
- [Result] Yavuz U, Sokucu S, Albayrak A, Ozturk K. Efficacy comparisons of the intraarticular steroidal agents in the patients with knee osteoarthritis. Rheumatol Int. 2012 Nov;32(11):3391-6. doi: 10.1007/s00296-011-2188-0. Epub 2011 Nov 5. PMID 22057944
- [Result] Wollstein R, Chaimsky G, Carlson L, Watson HK, Wollstein G, Saleh J. Evaluating short-term pain after steroid injection. Am J Orthop (Belle Mead NJ). 2007 Mar;36(3):128-31. PMID 17461394
- [Result] Kelly AM. The minimum clinically significant difference in visual analogue scale pain score does not differ with severity of pain. Emerg Med J. 2001 May;18(3):205-7. doi: 10.1136/emj.18.3.205. PMID 11354213
- [Result] Kuptniratsaikul V, Rattanachaiyanont M. Validation of a modified Thai version of the Western Ontario and McMaster (WOMAC) osteoarthritis index for knee osteoarthritis. Clin Rheumatol. 2007 Oct;26(10):1641-5. doi: 10.1007/s10067-007-0560-y. Epub 2007 Feb 20. PMID 17310271